CLINICAL TRIAL: NCT02313064
Title: A Two-Part, Double-Blind, Third Party Open (Sponsor), Dose-Rising, Placebo-Controlled and Open-Label Exploratory Food Effect Study of the Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of CXA-10 in Healthy Volunteers
Brief Title: Oral CXA-10 Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Complexa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CXA-10-201
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Kidney Injury
MeSH Terms: interventions — CXA-10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CXA-10 (Active Comparator): single dose of CXA-10 oral formulation
  Interventions: Drug: CXA-10
- CXA-10 placebo (Placebo Comparator): single oral doses of CXA-10 placebo
  Interventions: Drug: CXA-10 placebo

INTERVENTIONS:
Drug: CXA-10 — Part A has sequential single ascending doses will be administered in up to 5 cohorts of subjects. Each cohort of subjects will be randomized to receive a single dose of CXA-10 or placebo in, a fasted state. Part B has 2 periods and subjects will receive two doses of the selected dose of CXA-10.
  Arms: CXA-10
Drug: CXA-10 placebo
  Arms: CXA-10 placebo

SUMMARY:
This will be the first-in-human (FIH) study with the oral formulation of CXA-10. The main purpose of this trial is to demonstrate the safety, tolerability and pharmacokinetics (PK) of CXA-10 and its metabolite(s) administered as single ascending oral doses to healthy volunteers (Part A). The effects of food on the PK of CXA-10 will also be investigated (Part B).

DETAILED DESCRIPTION:
This will be the first-in-human (FIH) study with oral formulation of CXA-10. The main purpose of this trial is to demonstrate the safety, tolerability and pharmacokinetics (PK) of CXA-10 and its metabolite(s) administered as single ascending oral doses to healthy volunteers (Part A). The effects of food on the PK of CXA-10 will also be investigated (Part B). Part A of the study will be a single-center, randomized, double-blind, third party open (sponsor) placebo-controlled study. Sequential single ascending doses will be administered in up to 5 cohorts of subjects. Each cohort of subjects will be randomized to receive a single dose of CXA-10 or placebo in, a fasted state, as illustrated in the table below. Part B of the study will be a single-center, open-label, two-period study conducted in two cohorts of subjects as follows. The selected dose and the interval between Period 1 and Period 2 will be determined based on emerging PK data from Part A. The selected dose will be an intermediate dose level to avoid a food effect interaction that markedly enhances exposure. Subjects who participate in Part B of the study will receive two doses of CXA-10.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects and female subjects of non-child bearing potential between the ages of 18 and 50 years (inclusive)
2. Body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and a weight between 60 kg and 100 kg (inclusive)
3. In good general health as determined by a thorough medical history and physical examination, ECG, vital signs, and clinical laboratory evaluation. Results of clinical laboratory tests must be without clinically significant abnormalities, including hematology, clinical chemistry and urinalysis. Subjects with blood pressures less than 150/95 mmHg at screening may be enrolled
4. Subjects must have resting heart rates (HR) greater than or equal to 50 beats per minute at pre-dose
5. QTcF interval (Fredericia's correction factor) must be less than or equal to 430 msec for males and less than or equal to 450 msec for females at screening and pre-dose. Subjects with any other clinically relevant ECG parameter abnormality (e.g., PR interval, QRS deviation) or any clinically significant ECG abnormality will be excluded from the study. Subjects with a history of congenital long QT syndrome or in the subject's family will be excluded from the study (see Section 6.4)
6. Adequate venous access to allow for repeated blood sampling
7. Ability to comprehend and comply with procedures
8. Agree to commit to participate in the current protocol
9. Provide written informed consent prior to any study procedure being performed (all subjects should be able to understand the informed consent form and any other documents that subjects are required to read)

Exclusion Criteria:

1. Female subjects who are pregnant or lactating or who are trying to conceive
2. Females must not be of child bearing potential (defined as bilateral oophorectomy, hysterectomy, tubal ligation, or post-menopausal (amenorrhea for minimum of 1 year and post-menopausal status confirmed by follicle stimulating hormone (FSH) testing)). Female subjects unable to bear children (e.g. tubal ligation, hysterectomy, or post-menopausal) must have this documented in the case report form (CRF)
3. Female subjects with a positive urine β-human chorionic gonadotropin (β-hCG) test at screening or positive β-hCG urine at pre-dose
4. Any clinically relevant abnormality identified on the screening history, physical or laboratory examinations, or any other medical condition or circumstance making the volunteer unsuitable for participation in the study
5. Any clinical history of cardiovascular events, arrhythmias, fainting, palpitations, personal or family history of congenital prolonged QT syndromes or sudden unexpected death due to a cardiac reason
6. History of any primary malignancy, including a history of melanoma or suspicious undiagnosed skin lesions, with the exception of basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ or other malignancies curatively treated and with no evidence of disease for at least 5 years
7. History of regular alcohol consumption exceeding 14 units/week for women or 21 units/week for men (one unit equal to 125 mL of wine or 284 mL of beer or a single 25 mL measure of spirits) within 6 months of screening
8. History of smoking, including e-cigarettes, or use of nicotine-containing products within 1 month of screening
9. Treatment with any prescription or non-prescription drugs (including vitamins, herbal and dietary supplements) within 7 days or 5 half-lives, whichever is longer, prior to dosing and until collection of the final PK sample. Use of any drug including aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) must be avoided within 7 days prior to the first dose and during this study as it will interfere with the pharmacology of CXA-10. Use of high energy supplements or drinks (especially, those containing caffeine, protein supplements, and weight loss drugs) and smoking cessation products (gum, inhalers, patches, e cigarettes) will be prohibited

   -Only acetaminophen will be permitted at doses of 2 grams/day
10. Sitting blood pressure greater than 150 mmHg systolic and/or greater than 95 mmHg diastolic after 5 minutes rest (feet on floor, arm held at level of heart) at the screening visit
11. Resting heart rate greater than or equal to 100 beats per minute (BPM) after 5 minutes rest (as above) at the screening visit
12. Any abnormalities on 12-lead ECG at screening
13. Any clinically significant murmurs evident on auscultation of the heart (including evidence of mitral valve prolapse)
14. A positive urine drug screen for drugs of abuse, including alcohol or positive urine cotinine (greater than or equal to 300 ng/mL for cotinine) at the screening visit or at entry to the clinic (Note: urine cotinine required at screening visit only)
15. Treatment with any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the beginning of the screening period (this includes investigational formulations of marketed products, inhaled and topical drugs)
16. Blood collection of greater than 500 mL within 56 days prior to screening
17. Seropositive for human immunodeficiency virus (HIV) at screening
18. Positive for Hepatitis B virus surface antigen (HBsAg) or positive Hepatitis C virus antibody (HCV Ab) at screening
19. Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Serious and Non-Serious Adverse Events | First day of dosing through 30 days after the last dose
  Safety assessments will be performed prior to, during, and after dosing including a visit on Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blok, MD, Principal Investigator — Jasper Clinic, Michigan
Locations (1):
- Jasper Clinical Research & Development, Inc., Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No